CLINICAL TRIAL: NCT01108588
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-over Study Using Aspirin and Clopidogrel to Assess Reproducibility and Compare Platelet Function Assays
Brief Title: Reproducibility and Comparison of Platelet Function Assays With Aspirin and Clopidogrel (MK-0000-167)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-167; 167
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Aspirin - Clopidogrel - Placebo
  Interventions: Drug: Placebo (to match Aspirin); Drug: Aspirin; Drug: Clopidogrel; Drug: Comparator: Placebo (to match Clopidogrel)
- Sequence 2 (Experimental): Clopidogrel - Placebo - Aspirin
  Interventions: Drug: Placebo (to match Aspirin); Drug: Aspirin; Drug: Clopidogrel; Drug: Comparator: Placebo (to match Clopidogrel)
- Sequence 3 (Experimental): Placebo - Aspirin - Clopidogrel
  Interventions: Drug: Placebo (to match Aspirin); Drug: Aspirin; Drug: Clopidogrel; Drug: Comparator: Placebo (to match Clopidogrel)
- Sequence 4 (Experimental): Aspirin - Placebo - Clopidogrel
  Interventions: Drug: Placebo (to match Aspirin); Drug: Aspirin; Drug: Clopidogrel; Drug: Comparator: Placebo (to match Clopidogrel)
- Sequence 5 (Experimental): Clopidogrel - Aspirin - Placebo
  Interventions: Drug: Placebo (to match Aspirin); Drug: Aspirin; Drug: Clopidogrel; Drug: Comparator: Placebo (to match Clopidogrel)
- Sequence 6 (Experimental): Placebo - Clopidogrel - Aspirin
  Interventions: Drug: Placebo (to match Aspirin); Drug: Aspirin; Drug: Clopidogrel; Drug: Comparator: Placebo (to match Clopidogrel)

INTERVENTIONS:
Drug: Placebo (to match Aspirin) — Placebo grossly matched Aspirin 300 mg daily
Drug: Aspirin — Aspirin 300 mg daily
Drug: Clopidogrel — Clopidogrel 75 mg daily
Drug: Comparator: Placebo (to match Clopidogrel) — Placebo (grossly matched Clopidogrel 75 mg) daily

SUMMARY:
This study will evaluate whether the antiplatelet effects of Aspirin 300 mg daily and Clopidogrel 75 mg daily can be reproducibly measured using several point of care platelet function assays

ELIGIBILITY:
Inclusion Criteria:

* Subject has BMI (Body Mass Index) less than 32 kg/m^ 2
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 3 months
* Subject does not have a history of any bleeding disorder

Exclusion Criteria:

* Subject is a pregnant or nursing female
* Subject has a history of multiple and/or severe allergies to drugs or foods, or any history (personal or family) of bleeding disorders (including arterial bleeding, hemorrhage requiring transfusion or urgent intervention)
* Subject currently uses on a regular basis or has used aspirin or clopidogrel within 21 days prior to screening (including low-dose aspirin and pain relievers, cold, or sinus remedies containing aspirin)
* Subject currently uses on a regular basis or has used within 2 weeks prior to study start, any other prescription or nonprescription drugs, including NSAIDs such as ibuprofen, naproxen, COX-II inhibitors such as celecoxib or etoricoxib, other pain relievers, cold, or sinus remedies containing NSAIDs, and herbal remedies (e.g., St. John Wort)
* Subject anticipates needing during the study any prescription or nonprescription (including over the counter) preparation, including those that contain aspirin, ibuprofen, or any other NSAID or NSAID-containing product commonly found in pain relievers, cold or sinus remedies
* Subject has a history of skin conditions (such as dry skin, pruritus, rosacea, eczema) or has a sun burn at the time of screening and is unwilling to avoid excessive sun exposure for the duration of the study
* Subject regularly uses antacids or other OTC medications (4 or more times per month) for symptoms of dyspepsia or has a history of use of prescription ulcer medication such as H2 blockers (e.g., cimetidine, ranitidine, famotidine, nizatidine) or a proton pump inhibitor (omeprazole) within the last 5 years
* Subject has a history of poor wound healing or a tendency to form keloids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The effect size of light transmission platelet aggregation, bleeding time, and several point of care platelet function assays after 3 days of administration of study drug compared to placebo treatment. | Baseline and 3 days
The intra-subject coefficient of variation of each of the 3 platelet function devices | Baseline and 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Chen F, Maridakis V, O'neill EA, Beals C, Radziszewski W, de Lepeleire I, Van Dyck K, Depre M, Bolognese JA, de Hoon J, Jacquemin M. A randomized clinical trial comparing point-of-care platelet function assays and bleeding time in healthy subjects treated with aspirin or clopidogrel. Platelets. 2012;23(4):249-58. doi: 10.3109/09537104.2011.604806. Epub 2011 Sep 15. PMID 21919555